CLINICAL TRIAL: NCT07152613
Title: An Embedded Adaptive Randomized Controlled Trial of Corticosteroid Therapy for Pneumocystis Jirovecii Pneumonia (PJP) in Non-HIV Immunocompromised Patients
Brief Title: Corticosteroids for PJP in Non-HIV Immunocompromised Adults
Acronym: CAPSTONE-PJP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qingyuan Zhan (Other)
Responsible Party: Sponsor-Investigator, Qingyuan Zhan, Director, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-I2M-C&T-B-090B
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pneumocystis Jiroveci Pneumonia
Keywords: community-acquired pneumonia; Pneumocystis jiroveci; non-HIV; corticosteroids
MeSH Terms: conditions — Pneumonia, Pneumocystis; Community-Acquired Pneumonia | interventions — Sodium Chloride; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Placebo Comparator): Control Group
  Interventions: Drug: Saline (0.9%, sterile, for infusion)
- Low dose steroids (Experimental): Low dose steroids
  Interventions: Drug: Low Dose Corticosteroids
- Moderate dose steroids (Experimental): moderate dose steroids
  Interventions: Drug: Moderate dose corticosteroids

INTERVENTIONS:
Drug: Saline (0.9%, sterile, for infusion) — Saline for control
  Arms: Standard of Care
Drug: Low Dose Corticosteroids — Methylprednisolone 0.5mg/kg ivgtt qd
  Arms: Low dose steroids
Drug: Moderate dose corticosteroids — Methylprednisolone 1.0mg/kg ivgtt qd
  Arms: Moderate dose steroids

SUMMARY:
Pneumocystis jirovecii pneumonia (PJP) is one of the common severe complications in immunocompromised patients, with a reported mortality rate of 60-80%. Reducing mortality from PJP is crucial for improving outcomes in critically ill non-HIV immunocompromised patients and alleviating the burden on families and society. To address this medical challenge, our institution is conducting a study aimed at lowering PJP-related mortality. Specifically, we are performing an adaptive, randomized, open-label controlled trial in patients with severe PJP. The primary objective of this study is to scientifically evaluate the efficacy and safety of adjunctive corticosteroids at different dosages, in addition to early standard supportive care, for reducing mortality in severe PJP

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years.

Admission to the Intensive Care Unit (ICU).

Meeting the diagnostic criteria for community-acquired pneumonia (CAP).

Meeting at least one of the major diagnostic criteria for severe pneumonia:

(i) Requirement for endotracheal intubation and mechanical ventilation;

(ii) Septic shock requiring vasopressor therapy after adequate fluid resuscitation.

Or simultaneously fulfilling three of the minor criteria:

(i) Respiratory rate ≥ 30 breaths/min;

(ii) PaO₂/FiO₂ ≤ 250 mmHg;

(iii) Multilobar infiltrates;

(iv) Altered mental status and/or disorientation;

(v) Blood urea nitrogen ≥ 20 mg/dL (7.12 mmol/L);

(vi) Leukopenia (white blood cell count < 4 × 10⁹/L);

(vii) Thrombocytopenia (platelet count < 100 × 10⁹/L);

(viii) Hypothermia (core temperature < 36 °C);

(ix) Hypotension (systolic blood pressure < 90 mmHg) requiring aggressive fluid resuscitation.

Confirmed PJ etiology: at least one positive nucleic acid test (PCR) or next-generation sequencing (NGS) result for Pneumocystis jirovecii in respiratory specimens (respiratory secretions, throat swabs, or bronchoalveolar lavage fluid).

Severe community-acquired pneumonia (SCAP) patients admitted to the emergency department/ward/ICU due to respiratory failure within < 72 hours.

Signed informed consent.

Exclusion Criteria:

* Age < 18 years.
* Pregnant or breastfeeding women.
* HIV infection.
* No targeted PJP therapy administered or therapy not according to standard protocol.
* Diagnosis of PJP >7 days prior to MICU admission.
* Use of corticosteroids for PJP prior to MICU admission.
* Requirement for high-dose baseline corticosteroid therapy for other conditions (prednisone ≥ 0.5 mg/kg/day or equivalent).
* Any contraindication to corticosteroid use as judged by the investigator (e.g., severe concurrent infectious disease, severe gastrointestinal bleeding).
* Discharge or death within 48 hours after intervention.
* Participation in other clinical studies or refusal to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
28-days all cause mortality | 28 days from inclusion
  28-days all cause mortality

IPD SHARING:
Plan to Share IPD: Undecided